CLINICAL TRIAL: NCT02124733
Title: Simultaneous Incubation/Illumination Versus Short Aminolevulinate Preincubation for Painless Photodynamic Therapy of Actinic Keratoses
Brief Title: Protocols for Painless Photodynamic Therapy (PDT) of Actinic Keratoses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Edward Maytin, MD, PhD, MD, PhD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-374
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Actinic Keratoses; AK; PDT; Photodynamic Therapy; Blue Light Therapy; ALA; aminolevulinic acid; Levulan
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Patients with actinic keratosis of the face/scalp were enrolled for an intrapatient comparative study of two different regimens for delivering ALA-based PDT treatment. In this contralateral/bilateral study design, each patient served as his/her own control. One side of the face or scalp (Side B), the traditional control regimen of PDT was given (1 h topical drug then 16 min 40 sec of blue light). On the test side (Side A), we administered a new regimen; topical drug was applied and then the blue light immediately started. Three groups of patients (Study arms) had different times of exposure (either 30 min, 45 min, or 60 min). For all patients, the post-treatment course was compared for Sides A vs. B. The primary endpoints were pain during illumination, and lesion clearance at 3 months post-therapy.
Who Masked: Outcomes Assessor
Masking Description: Evaluator assesses photographs without prior knowledge of intervention
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: 30 minutes (Active Comparator): The first 4 patients enrolled will be considered Group 1, and will receive 30 min of Aminolevulinic acid based photodynamic therapy to Side A. They will be evaluated in terms of erythema immediately post-PDT (Day 1) and on Day 4 . If there is no clinical reaction on Side A after 2 patients, then the dose will be advanced to the next Group. If the post-PDT reaction (erythema at Day 4) on Side A equals or exceeds the reaction on Side B in the majority of the first 4 patients, then the dose will not be escalated and recruitment will continue until 15 patients have been treated (thereby completing the study). If the post-PDT reaction on Side A is less than the reaction on Side B in the majority of the 4 patients, then the protocol will advance to Group 2
  Interventions: Procedure: Aminolevulinic acid based photodynamic therapy
- Group 2: 45 minutes (Active Comparator): Patients in this group will receive 45 min of Aminolevulinic acid based photodynamic therapy to Side A. They will be evaluated for erythema response immediately post-PDT and at Day 4. If there is no clinical reaction on Side A after 2 patients, then the dose will be advanced to the next Group. If the post-PDT reaction (erythema at Day 4) on Side A equals or exceeds the reaction on Side B in the majority of the first 4 patients, then the dose will not be escalated and recruitment will continue until 15 patients have been treated (thereby completing the study). If the post-PDT reaction on Side A is less than the reaction on Side B in the majority of the 4 patients, then the protocol will advance to Group 3.
  Interventions: Procedure: Aminolevulinic acid based photodynamic therapy
- Group 3: 60 minutes (Active Comparator): Patients in this group will receive 60 min of Aminolevulinic acid based photodynamic therapy to Side A. They will be evaluated for erythema responses immediately post-PDT and at Day 4. If the post-PDT reaction on Side A equals or exceeds the reaction on Side B in the majority of the first 4 patients, then the dose will not be escalated and recruitment will continue until 15 patients have been treated (thereby completing the study). If the post-PDT reaction on Side A is less than the reaction on Side B in the majority of patients, then the protocol will terminate after 15 patients (total for all groups) have been treated.
  Interventions: Procedure: Aminolevulinic acid based photodynamic therapy

INTERVENTIONS:
Procedure: Aminolevulinic acid based photodynamic therapy — The PDT treatments will be done in two stages. ALA (Levulan® Kerastick™) will be applied to the entire treatment area, and then the longer light exposure (lasting up to 1 hr) will be performed on one-half of the treatment area (Side A). After that, a shorter (16 min 40 sec) light exposure will be done on the other half (Side B).
  Other Names: Levulan® Kerastick™; Blu-U

SUMMARY:
This study is being done to compare a new, continuous illumination regimen of ALA-PDT (Aminolevulinate-Photodynamic Therapy) to a conventional regimen for treatment of actinic keratoses. The hypothesis is that the continuous illumination approach will be less painful, but equally efficacious, as the old regimen.

DETAILED DESCRIPTION:
This study is being done to compare a modified version of the standard ALA-PDT (Aminolevulinate-Photodynamic Therapy) treatment of actinic keratoses, to a modified version in which light exposure begins immediately after application of the Levulan. We hypothesize that this will yield a therapeutic efficacy equivalent to the standard ALA-PDT regimen, but will cause less pain during the light exposure. The study employs a bilateral design in which the left versus right sides of the treatment area are compared in the exact same patient. There are 3 arms of the study, each having a different time duration of light exposure in the modified regimen to determine which one is most efficacious

ELIGIBILITY:
Inclusion Criteria:

* Males or females, at least 18 years of age
* Non-hyperkeratotic actinic keratoses, at least 6 in number (3 on each side of scalp, face or upper extremities)

Exclusion Criteria:

* patient is currently pregnant or are planning to conceive during the course of the study period
* patient is using topical therapy or other treatment for these actinic keratoses
* patient has a known hypersensitivity to 5-aminolevulinic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
AK clearance | at 3 months post-treatment
  The primary endpoint is treatment efficacy (AK lesion clearance at 3 months). The specific aim of this study is to establish proof-of-principle for the concept that a long delivery period of blue light from the Blu-U device, using the standard fluence rate but starting only 15 min after the application of Levulan and lasting 1 hour (fluence of 360 J/cm2), can provide a clearance rate of AK lesions comparable to a standard regimen of Blu-U light (fluence of 10 J/cm2) beginning 1 hr after LevulanTM application.

SECONDARY OUTCOMES:
Pain during illumination | During treatment through post-treatment Day4
  The secondary endpoint is pain during illumination. The hypothesis is that efficacy at 3 months will be statistically equivalent with the two approaches, but pain will be significantly less with the continuous treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Maytin, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States